CLINICAL TRIAL: NCT00975286
Title: A Randomized, Placebo-controlled, 2-arm Parallel-group, Multicenter Study With a 24-week Double-blind Treatment Period Assessing the Efficacy and Safety of Lixisenatide in Patients With Type 2 Diabetes Insufficiently Controlled With Insulin Glargine and Metformin
Brief Title: 24-week Treatment With Lixisenatide in Type 2 Diabetes Insufficiently Controlled With Metformin and Insulin Glargine
Acronym: GetGoal-Duo1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC10781; EudraCT : 2008-007335-40
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Insulin Glargine; Metformin; 2,4-thiazolidinedione

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lixisenatide (Experimental): 2-step initiation regimen of lixisenatide: 10 microgram (mcg) once daily (QD) for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Insulin glargine; Device: Pen auto-injector; Drug: Metformin; Drug: Thiazolidinedione (TZD)
- Placebo (Placebo Comparator): 2-step initiation regimen of volume matching placebo: 10 mcg QD for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
  Interventions: Drug: Placebo; Drug: Insulin glargine; Device: Pen auto-injector; Drug: Metformin; Drug: Thiazolidinedione (TZD)

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Lixisenatide
Drug: Placebo — Self administered by subcutaneous injections once daily within the hour preceding breakfast.
  Arms: Placebo
Drug: Insulin glargine — Dose to be adjusted to maintain a fasting SMPG between 100 and 80 mg/dL (5.6 and 4.4 mmol/L), inclusive.
  Other Names: Lantus®
Device: Pen auto-injector — Lantus® SoloStar® OptiClik®
Drug: Metformin — Metformin to be continued at stable dose (at least 1.5 gram per day) up to Week 24.
Drug: Thiazolidinedione (TZD) — TZD (either rosiglitazone or pioglitazone) if given, to be continued at stable dose up to Week 24.

SUMMARY:
The purpose of the study is to evaluate the benefits and risks of lixisenatide (AVE0010), in comparison to placebo, as an add-on treatment to insulin glargine and metformin with or without thiazolidinediones (TZDs), over a period of 24 weeks of treatment.

The primary objective is to assess the effects of lixisenatide in comparison to placebo, when added to insulin glargine and metformin, on glycemic control in terms of glycosylated hemoglobin (HbA1c) reduction (absolute change) at Week 24.

The secondary objectives are to assess the effects of lixisenatide on the percentage of patients reaching HbA1c less than (<) 7 percent (%) and less than or equal to (<=) 6.5%, plasma glucose (fasting, postprandial during a standardized meal challenge test, 7-point self monitored profiles), body weight, insulin glargine doses, to evaluate safety and tolerability (including anti-lixisenatide antibody assessment), and to assess the impact on treatment satisfaction using the Diabetes Treatment Satisfaction Questionnaire (state) (DTSQs) in the participating countries where it is validated.

DETAILED DESCRIPTION:
The study comprises 3 periods:

* An up to 14-week screening period, which includes an up to 2-week screening phase and a 12-week run-in phase with introduction and titration of insulin glargine on top of metformin +/-TZDs.
* At the end of the run-in phase, patients whose HbA1c (centralized assay) is greater than or equal to (>=) 7% and less than or equal to (<=) 9% and whose mean fasting self-monitored plasma glucose (SMPG) calculated from the self measurements for the 7 days prior to Visit 12 (Week -1) is <=140 milligram per deciliter (mg/dL) (7.8 millimole per liter [mmol/L]), would enter a 24-week double-blind randomized treatment period comparing lixisenatide to placebo (on top of insulin glargine + metformin +/- TZDs).
* A 3-day safety follow up period.

Maximum duration is of 39 weeks +/- 7 days.

ELIGIBILITY:
Inclusion criteria:

- Type 2 diabetes mellitus, diagnosed for at least 1 year before screening visit, insufficiently controlled with insulin glargine and metformin

Exclusion criteria:

* HbA1c <7% or greater than (>)10% at screening
* At the time of screening age < legal age of majority
* Pregnant or breastfeeding women or women of childbearing potential with no effective contraceptive method
* Type 1 diabetes mellitus
* Metformin not at a stable dose of at least 1.5 gram per day for at least 3 months prior to the screening visit
* Use of oral or injectable antidiabetic or hypoglycemic agents other than metformin, sulfonylurea (SU) and TZDs (for example, alpha glucosidase inhibitor, other glucagon like peptide-1 [GLP-1] receptor agonists, dipeptidyl peptidase-IV [DPP-IV] inhibitors, insulin etc.) within 3 months prior to the time of screening, use of weight loss drugs if not at a stable dose for at least 3 months prior to the screening visit
* History of hypoglycemia unawareness
* Body Mass Index (BMI) less than or equal to (<=) 20 kilogram per square meter (kg/m^2)
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease, personal or family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (for example, multiple endocrine neoplasia syndromes)
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening
* Hemoglobinopathy or hemolytic anemia, blood or plasma products transfusion within 3 months prior to the time of screening
* Within the last 6 months prior to screening: history of myocardial infarction, stroke, or heart failure requiring hospitalization
* Known history of drug or alcohol abuse within 6 months prior to the time of screening
* Any clinically significant abnormality identified on physical examination, laboratory tests, electrocardiogram or vital signs at the time of screening that in the judgment of the Investigator or any sub investigator precludes safe completion of the study or constrains efficacy assessment such as active malignant tumor or other major systemic diseases, presence of clinically significant diabetic retinopathy or presence of macular edema likely to require laser treatment within the study period
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting systolic or diastolic blood pressure >180 millimeter of mercury (mmHg) or >110 mmHg, respectively
* Laboratory findings at the time of screening: amylase and/or lipase, alanine aminotransferase >3 times upper limit of the normal (ULN) laboratory range; total bilirubin: >1.5 times ULN (except in case of Gilbert's syndrome); hemoglobin <11 gram/deciliter and/or neutrophils <1500 per cubic millimeter (mm^3) and/or platelets <100 000/mm^3; positive test for Hepatitis B surface antigen and/or Hepatitis C antibody, positive serum pregnancy test in females of childbearing potential; and calcitonin >=20 picogram per milliliter (pg/mL) (5.9 picomole per milliliter [pmol/L])
* Patients who are considered by the Investigator or any sub investigator as inappropriate for this study for any reason (for example, impossibility to meet specific protocol requirements, such as scheduled visits, being able to do self-injections, likelihood of requiring treatment during the screening phase and treatment phase with drugs not permitted by the clinical study protocol, patient being investigator or any sub investigator, pharmacist, study coordinator, other study staff or relative thereof directly involved in the conduct of the protocol etc.)
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for one week or more within 3 months prior to the time of screening
* Use of any investigational drug within 3 months prior to screening
* Renal impairment defined with serum creatinine > 1.4 mg/dL in women and > 1.5 mg/dL in men
* History of hypersensitivity to insulin glargine or to any of the excipients
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to): gastroparesis, unstable (that is, worsening) and not controlled (that is, prolonged nausea and vomiting) gastroesophageal reflux disease requiring medical treatment, within 6 months prior to the time of screening
* Any previous treatment with lixisenatide (for example, participation in a previous study with lixisenatide)
* Allergic reaction to any GLP-1 receptor agonist in the past (for example, exenatide, liraglutide) or to metacresol
* Additional exclusion criteria during or at the end of the run-in phase before randomization: informed consent withdrawal (patient who was not willing to continue or failed to return), mean fasting SMPG calculated from the self-measurements for the 7 days prior to Visit 12 (Week -1) was >140 mg/dL (7.8 mmol/L) and HbA1c measured at Visit 12 (Week -1) is <7% or >9%, amylase and/or lipase > 3 times the ULN at Visit 12 (Week -1), patients with fasting plasma glucose (FPG) above the threshold value described for rescue (that is, FPG >240 mg/dL [13.3 mmol/L]), patients with any adverse event, which, by the judgment of the Investigator precludes the inclusion in the double-blind randomized treatment phase, and lack of compliance to protocol or to insulin glargine treatment during the run-in phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Operations, Study Director — Sanofi
Locations (140):
- United States (23):
  - Sanofi-Aventis Investigational Site Number 840223, Mesa, Arizona
  - Sanofi-Aventis Investigational Site Number 840206, Hot Springs, Arkansas
  - Sanofi-Aventis Investigational Site Number 840201, Little Rock, Arkansas
  - Sanofi-Aventis Investigational Site Number 840212, Mountain Home, Arkansas
  - Sanofi-Aventis Investigational Site Number 840215, Concord, California
  - Sanofi-Aventis Investigational Site Number 840214, Greenbrae, California
  - Sanofi-Aventis Investigational Site Number 840221, Orlando, Florida
  - Sanofi-Aventis Investigational Site Number 840211, Baton Rouge, Louisiana
  - Sanofi-Aventis Investigational Site Number 840230, Hyattsville, Maryland
  - Sanofi-Aventis Investigational Site Number 840209, Rockville, Maryland
  - Sanofi-Aventis Investigational Site Number 840219, Brighton, Michigan
  - Sanofi-Aventis Investigational Site Number 840231, Sea Girt, New Jersey
  - Sanofi-Aventis Investigational Site Number 840208, Fargo, North Dakota
  - Sanofi-Aventis Investigational Site Number 840225, Mentor, Ohio
  - Sanofi-Aventis Investigational Site Number 840222, Portland, Oregon
  - Sanofi-Aventis Investigational Site Number 840202, Philadelphia, Pennsylvania
  - Sanofi-Aventis Investigational Site Number 840229, Bristol, Tennessee
  - Sanofi-Aventis Investigational Site Number 840205, Germantown, Tennessee
  - Sanofi-Aventis Investigational Site Number 840210, Dallas, Texas
  - Sanofi-Aventis Investigational Site Number 840217, Houston, Texas
  - Sanofi-Aventis Investigational Site Number 840228, Houston, Texas
  - Sanofi-Aventis Investigational Site Number 840213, Plano, Texas
  - Sanofi-Aventis Investigational Site Number 840227, Norfolk, Virginia
- Argentina (7):
  - Sanofi-Aventis Investigational Site Number 032204, Buenos Aires
  - Sanofi-Aventis Investigational Site Number 032205, Capital Federal
  - Sanofi-Aventis Investigational Site Number 032201, Capital Federal
  - Sanofi-Aventis Investigational Site Number 032209, Capital Federal
  - Sanofi-Aventis Investigational Site Number 032211, Corrientes
  - Sanofi-Aventis Investigational Site Number 032202, Paraná
  - Sanofi-Aventis Investigational Site Number 032203, Rosario
- Brazil (4):
  - Sanofi-Aventis Investigational Site Number 076207, Belém
  - Sanofi-Aventis Investigational Site Number 076202, Brasília
  - Sanofi-Aventis Investigational Site Number 076205, Porto Alegre
  - Sanofi-Aventis Investigational Site Number 076204, São Paulo
- Canada (11):
  - Sanofi-Aventis Investigational Site Number 124219, Brampton
  - Sanofi-Aventis Investigational Site Number 124213, Chatham
  - Sanofi-Aventis Investigational Site Number 124208, Chilliwack
  - Sanofi-Aventis Investigational Site Number 124215, Etobicoke
  - Sanofi-Aventis Investigational Site Number 124205, Québec
  - Sanofi-Aventis Investigational Site Number 124202, Red Deer
  - Sanofi-Aventis Investigational Site Number 124218, Thornhill
  - Sanofi-Aventis Investigational Site Number 124201, Toronto
  - Sanofi-Aventis Investigational Site Number 124207, Toronto
  - Sanofi-Aventis Investigational Site Number 124209, Victoria
  - Sanofi-Aventis Investigational Site Number 124217, Winnipeg
- Chile (6):
  - Sanofi-Aventis Investigational Site Number 152202, Santiago
  - Sanofi-Aventis Investigational Site Number 152203, Santiago
  - Sanofi-Aventis Investigational Site Number 152206, Santiago
  - Sanofi-Aventis Investigational Site Number 152204, Santiago
  - Sanofi-Aventis Investigational Site Number 152205, Santiago
  - Sanofi-Aventis Investigational Site Number 152201, Santiago
- Colombia (3):
  - Sanofi-Aventis Investigational Site Number 170204, Barranquilla
  - Sanofi-Aventis Investigational Site Number 170201, Bogotá
  - Sanofi-Aventis Investigational Site Number 170202, Bogotá
- Czechia (2):
  - Sanofi-Aventis Investigational Site Number 203202, Hradec Králové
  - Sanofi-Aventis Investigational Site Number 203204, Prague
- Denmark (3):
  - Sanofi-Aventis Investigational Site Number 208202, Frederiksberg
  - Sanofi-Aventis Investigational Site Number 208201, København NV
  - Sanofi-Aventis Investigational Site Number 208205, Slagelse
- Estonia (4):
  - Sanofi-Aventis Investigational Site Number 233201, Pärnu
  - Sanofi-Aventis Investigational Site Number 233203, Tallinn
  - Sanofi-Aventis Investigational Site Number 233204, Tartu
  - Sanofi-Aventis Investigational Site Number 233202, Viljandimaa
- France (5):
  - Sanofi-Aventis Investigational Site Number 250204, Amiens
  - Sanofi-Aventis Investigational Site Number 250206, La Rochelle
  - Sanofi-Aventis Investigational Site Number 250203, Le Creusot
  - Sanofi-Aventis Investigational Site Number 250201, Nantes
  - Sanofi-Aventis Investigational Site Number 250202, Pierre-Bénite
- Germany (3):
  - Sanofi-Aventis Investigational Site Number 276201, Dresden
  - Sanofi-Aventis Investigational Site Number 276202, Mainz
  - Sanofi-Aventis Investigational Site Number 276204, Saint Ingbert-Oberwürzbach
- Hungary (7):
  - Sanofi-Aventis Investigational Site Number 348205, Balatonfüred
  - Sanofi-Aventis Investigational Site Number 348202, Budapest
  - Sanofi-Aventis Investigational Site Number 348207, Budapest
  - Sanofi-Aventis Investigational Site Number 348204, Debrecen
  - Sanofi-Aventis Investigational Site Number 348206, Gyula
  - Sanofi-Aventis Investigational Site Number 348203, Szeged
  - Sanofi-Aventis Investigational Site Number 348201, Zalaegerszeg
- India (10):
  - Sanofi-Aventis Investigational Site Number 356210, Ahmedabad
  - Sanofi-Aventis Investigational Site Number 356206, Bangalore
  - Sanofi-Aventis Investigational Site Number 356204, Bangalore
  - Sanofi-Aventis Investigational Site Number 356202, Bangalore
  - Sanofi-Aventis Investigational Site Number 356201, Belagavi
  - Sanofi-Aventis Investigational Site Number 356205, Chennai
  - Sanofi-Aventis Investigational Site Number 356208, Indore
  - Sanofi-Aventis Investigational Site Number 356203, Karnāl
  - Sanofi-Aventis Investigational Site Number 356207, Kochi
  - Sanofi-Aventis Investigational Site Number 356209, Nagpur
- Israel (4):
  - Sanofi-Aventis Investigational Site Number 376202, Haifa
  - Sanofi-Aventis Investigational Site Number 376201, Holon
  - Sanofi-Aventis Investigational Site Number 376204, Kfar Saba
  - Sanofi-Aventis Investigational Site Number 376203, Tel Litwinsky
- Italy (2):
  - Sanofi-Aventis Investigational Site Number 380201, Milan
  - Sanofi-Aventis Investigational Site Number 380202, Perugia
- Malaysia (2):
  - Sanofi-Aventis Investigational Site Number 458203, Kelantan
  - Sanofi-Aventis Investigational Site Number 458202, Kuala Lumpur
- Mexico (5):
  - Sanofi-Aventis Investigational Site Number 484201, Cuernavaca
  - Sanofi-Aventis Investigational Site Number 484204, Durango
  - Sanofi-Aventis Investigational Site Number 484203, Guadalajara
  - Sanofi-Aventis Investigational Site Number 484206, México
  - Sanofi-Aventis Investigational Site Number 484205, Tlalnepantla
- Netherlands (3):
  - Sanofi-Aventis Investigational Site Number 528203, Amsterdam
  - Sanofi-Aventis Investigational Site Number 528202, Groningen
  - Sanofi-Aventis Investigational Site Number 528204, Zwijndrecht
- Poland (7):
  - Sanofi-Aventis Investigational Site Number 616202, Krakow
  - Sanofi-Aventis Investigational Site Number 616208, Lubin
  - Sanofi-Aventis Investigational Site Number 616207, Puławy
  - Sanofi-Aventis Investigational Site Number 616206, Płock
  - Sanofi-Aventis Investigational Site Number 616205, Sopot
  - Sanofi-Aventis Investigational Site Number 616201, Szczecin
  - Sanofi-Aventis Investigational Site Number 616203, Zabrze
- Puerto Rico (2):
  - Sanofi-Aventis Investigational Site Number 840226, Ponce
  - Sanofi-Aventis Investigational Site Number 840216, San Juan
- Romania (8):
  - Sanofi-Aventis Investigational Site Number 642204, Brasov
  - Sanofi-Aventis Investigational Site Number 642208, Bucharest
  - Sanofi-Aventis Investigational Site Number 642205, Deva
  - Sanofi-Aventis Investigational Site Number 642203, Iași
  - Sanofi-Aventis Investigational Site Number 642202, Oradea
  - Sanofi-Aventis Investigational Site Number 642206, Târgu Mureş
  - Sanofi-Aventis Investigational Site Number 642207, Timișoara
  - Sanofi-Aventis Investigational Site Number 642201, Timișoara
- Russia (2):
  - Sanofi-Aventis Investigational Site Number 643202, Saint Petersburg
  - Sanofi-Aventis Investigational Site Number 643203, Saratov
- South Africa (3):
  - Sanofi-Aventis Investigational Site Number 710202, Cape Town
  - Sanofi-Aventis Investigational Site Number 710201, Durban
  - Sanofi-Aventis Investigational Site Number 710203, Pretoria
- Sweden (5):
  - Sanofi-Aventis Investigational Site Number 752204, Gothenburg
  - Sanofi-Aventis Investigational Site Number 752203, Härnösand
  - Sanofi-Aventis Investigational Site Number 752205, Luleå
  - Sanofi-Aventis Investigational Site Number 752202, Malmo
  - Sanofi-Aventis Investigational Site Number 752201, Stockholm
- Taiwan (4):
  - Sanofi-Aventis Investigational Site Number 158204, Changhua
  - Sanofi-Aventis Investigational Site Number 158203, Taichung
  - Sanofi-Aventis Investigational Site Number 158201, Taichung R.o.c.
  - Sanofi-Aventis Investigational Site Number 158202, Tainan Hsien
- Ukraine (5):
  - Sanofi-Aventis Investigational Site Number 804203, Chernivtsi
  - Sanofi-Aventis Investigational Site Number 804201, Kiev
  - Sanofi-Aventis Investigational Site Number 804205, Kyiv
  - Sanofi-Aventis Investigational Site Number 804202, Kyiv
  - Sanofi-Aventis Investigational Site Number 804204, Vinnytsia

REFERENCES:
- [Result] Riddle MC, Forst T, Aronson R, Sauque-Reyna L, Souhami E, Silvestre L, Ping L, Rosenstock J. Adding once-daily lixisenatide for type 2 diabetes inadequately controlled with newly initiated and continuously titrated basal insulin glargine: a 24-week, randomized, placebo-controlled study (GetGoal-Duo 1). Diabetes Care. 2013 Sep;36(9):2497-503. doi: 10.2337/dc12-2462. Epub 2013 Apr 5. PMID 23564915
- [Derived] Yao J, Zhang M, Zhang X, Zhang J. Impact of Type 2 Diabetes Duration on the Efficacy and Safety of Add-on Lixisenatide in Asian Individuals Receiving Basal Insulin: A Pooled Analysis. Diabetes Ther. 2023 Apr;14(4):653-669. doi: 10.1007/s13300-023-01369-6. Epub 2023 Feb 21. PMID 36809495
- [Derived] Davidson JA, Stager W, Paranjape S, Berria R, Leiter LA. Achieving postprandial glucose control with lixisenatide improves glycemic control in patients with type 2 diabetes on basal insulin: a post-hoc analysis of pooled data. Clin Diabetes Endocrinol. 2020 Jan 14;6:2. doi: 10.1186/s40842-019-0088-5. eCollection 2020. PMID 31956422
- [Derived] Rosenstock J, Handelsman Y, Vidal J, Ampudia Blasco FJ, Giorgino F, Liu M, Perfetti R, Meier JJ. Propensity-score-matched comparative analyses of simultaneously administered fixed-ratio insulin glargine 100 U and lixisenatide (iGlarLixi) vs sequential administration of insulin glargine and lixisenatide in uncontrolled type 2 diabetes. Diabetes Obes Metab. 2018 Dec;20(12):2821-2829. doi: 10.1111/dom.13462. Epub 2018 Aug 13. PMID 29974618
- [Derived] Charbonnel B, Bertolini M, Tinahones FJ, Domingo MP, Davies M. Lixisenatide plus basal insulin in patients with type 2 diabetes mellitus: a meta-analysis. J Diabetes Complications. 2014 Nov-Dec;28(6):880-6. doi: 10.1016/j.jdiacomp.2014.07.007. Epub 2014 Jul 18. PMID 25130920
- [Derived] Riddle MC, Aronson R, Home P, Marre M, Niemoeller E, Miossec P, Ping L, Ye J, Rosenstock J. Adding once-daily lixisenatide for type 2 diabetes inadequately controlled by established basal insulin: a 24-week, randomized, placebo-controlled comparison (GetGoal-L). Diabetes Care. 2013 Sep;36(9):2489-96. doi: 10.2337/dc12-2454. Epub 2013 Apr 29. PMID 23628617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 140 centers in 25 countries between October 13, 2009 and August 01, 2011.
Pre-assignment Details: A total of 1470 patients were screened of which 1024 were screen or run-in failures; main reason for screen failure was glycosylated hemoglobin (HbA1c) values being out of the defined protocol range (greater than or equal to 7% and less than or equal to 9%). A total of 446 patients were randomized.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 microgram (mcg) once daily (QD) subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
- Lixisenatide: 2-step initiation regimen of lixisenatide: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
Period: Overall Study
Arm/Group | Placebo | Lixisenatide
Started | 223 (Randomized.) | 223
Safety Population | 223 (All patients who were exposed to at least 1 dose, regardless of amount of treatment administered.) | 223
Modified Intent-to-Treat(mITT)Population | 223 (All patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment.) | 223
Completed | 211 | 194
Not Completed | 12 | 29
Not completed — Adverse Event | 9 | 19
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Familial and Personal Reasons | 2 | 2
Not completed — Poor Compliance to Protocol | 0 | 2
Not completed — Sponsor Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo: 10 mcg QD subcutaneously for 1 week, followed by 15 mcg QD for 1 week, then 20 mcg QD up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lixisenatide | Total
Number analyzed (Participants) | 223 | 223 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at screening is reported.
  years | 56.1 (10.2) | 56.4 (9.7) | 56.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 114 | 224
  Male | 113 | 109 | 222
Race/Ethnicity, Customized [Number; unit: participants]
  Race: Caucasian/White | 167 | 165 | 332
  Race: Black | 11 | 9 | 20
  Race: Asian/Oriental | 43 | 44 | 87
  Race: Other | 2 | 5 | 7
  Ethnicity: Hispanic | 49 | 52 | 101
  Ethnicity: Non Hispanic | 174 | 171 | 345
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of hemoglobin] | 7.60 (0.54) | 7.56 (0.55) | 7.58 (0.54)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 6.70 (1.97) | 6.55 (1.72) | 6.62 (1.85)
2-Hour Postprandial Plasma Glucose (PPG) [Mean (Standard Deviation); unit: mmol/L] — The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Number of patients evaluable for this Baseline characteristic were 221 and 219 for Placebo and Lixisenatide arm, respectively.
  mmol/L | 12.79 (3.69) | 12.90 (3.94) | 12.85 (3.81)
Glucose Excursion [Mean (Standard Deviation); unit: mmol/L] — Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the meal test, before study drug administration. Number of patients evaluable for this Baseline characteristic were 221 and 219 for Placebo and Lixisenatide arm, respectively.
  mmol/L | 6.33 (3.54) | 6.24 (4.35) | 6.29 (3.96)
Average 7-Point Self Monitored Plasma Glucose (SMPG) [Mean (Standard Deviation); unit: mmol/L] — Patients recorded a 7-point plasma glucose profile before and 2 hours after each meal and at bedtime once in a week and the average value for the 7-time points was calculated. Number of patients evaluable for this Baseline characteristic were 221 and 221 for Placebo and Lixisenatide arm, respectively.
  mmol/L | 8.26 (1.52) | 8.20 (1.47) | 8.23 (1.49)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 86.75 (20.41) | 87.31 (21.76) | 87.03 (21.07)
Average Insulin Glargine Daily Dose [Mean (Standard Deviation); unit: units per day] — Insulin glargine average daily dose at Baseline is the average daily dose for the week prior to Visit 12 (Week -1).
  units per day | 44.24 (19.86) | 43.44 (18.84) | 43.84 (19.34)
Treatment Satisfaction Score (Diabetes Treatment Satisfaction Questionnaire [DTSQ]) [Mean (Standard Deviation); unit: units on a scale] — DTSQ: 8-item questionnaire to assess treatment satisfaction and patient perception of hyper and hypoglycemia. Each question (Q) scored on a Likert scale from 0 (worst case) to 6 (best case) except Q2 and 3 where 0 (best case) to 6 (worst case). Six items (Q1 and 4-8) measured treatment satisfaction and were summed to calculate treatment satisfaction score which ranged from 0 (very dissatisfied) to 36 (very satisfied). Two items (Q2 and 3), which were not included, measured perceived hyperglycemia and hypoglycemia, respectively and lower score represented good perceived blood glucose control.
  units on a scale | 31.5 (5.1) | 31.7 (4.5) | 31.6 (4.8)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Duration of diabetes at screening is reported.
  years | 8.72 (5.82) | 9.62 (6.03) | 9.17 (5.94)
Metformin Daily Dose [Mean (Standard Deviation); unit: milligram (mg) per day] | 2058.1 (430.6) | 2039.2 (405.3) | 2048.7 (417.8)
Number of Patients With Thiazolidinedione (TZD) use at Baseline [Number; unit: participants]
  Yes | 27 | 27 | 54
  No | 196 | 196 | 392
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI was calculated by dividing body weight by the height squared.
  kilogram per square meter (kg/m^2) | 31.65 (6.01) | 31.99 (6.63) | 31.82 (6.32)
Number of Patients With Categorical BMI [Number; unit: participants]
  Less than 30 | 103 | 103 | 206
  Greater than or equal to 30 | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Absolute change = HbA1c value at Week 24 minus HbA1c value at baseline. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 14 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population:all randomized patients who received at least 1 dose;had baseline,at least 1 post-baseline efficacy assessment, irrespective of compliance with study protocol/procedures. Number of patients analyzed=patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period. Last observation carried forward used.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Groups:
- Placebo: 2-step initiation regimen of volume matching placebo.
- Lixisenatide: 2-step initiation regimen of lixisenatide.
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 221 | 215
percentage of hemoglobin | -0.40 (0.092) | -0.71 (0.091)
Statistical Analysis 1: Comparison: Placebo vs Lixisenatide; To detect a difference of 0.5% (or 0.4%) in change from baseline to Week 24 in HbA1c between lixisenatide and placebo, 225 patients in each arm would provide a power of 98% (or 90%) assuming common standard deviation of 1.3% with a 2-sided test at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANCOVA — Statistical testing: 2-sided at significance level=0.05. Analysis of covariance (ANCOVA) included treatment arms; randomization strata of Week -1 HbA1c (<8.0,>=8.0%) and TZD use (yes/no); country as fixed effects; baseline HbA1c as covariate; [Least squares (LS) mean difference = -0.32, 95% CI 2-sided [-0.463 to -0.171], Standard Error of Mean 0.074

2. Secondary Outcome: Change From Baseline in 2-Hour Postprandial Plasma Glucose (PPG) at Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline 2-hour PPG assessment during on-treatment period. Missing data was imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 204 | 194
mmol/L | 0.08 (0.481) | -3.09 (0.482)

3. Secondary Outcome: Change From Baseline in Glucose Excursion at Week 24
Description: Glucose excursion = 2-hour PPG minus plasma glucose 30 minutes prior to the standardized meal test, before study drug administration. Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline glucose excursion assessment during on-treatment period. Missing data was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 204 | 194
mmol/L | -0.33 (0.461) | -3.42 (0.462)

4. Secondary Outcome: Change From Baseline in Average 7-Point Self Monitored Plasma Glucose (SMPG) Profile at Week 24
Description: Patients recorded a 7-point plasma glucose profile measured before and 2 hours after each meal and at bedtime once in a week and the average value for the 7-time points was calculated. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline average 7-point SMPG assessment during on-treatment period. Missing data was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 214 | 210
mmol/L | -0.08 (0.179) | -0.47 (0.178)

5. Secondary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period. Missing data was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 220 | 217
kilogram | 1.16 (0.330) | 0.28 (0.331)

6. Secondary Outcome: Change From Baseline in Average Insulin Glargine Daily Dose at Week 24
Description: Change was calculated by subtracting the baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to the last dosing day of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline insulin glargine dose assessment during on-treatment period. Missing data was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units per day
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 223 | 222
units per day | 5.34 (1.256) | 3.10 (1.260)

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 1 day after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline FPG assessment during on-treatment period. Missing data was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 220 | 214
mmol/L | 0.46 (0.214) | 0.34 (0.213)

8. Other Pre Specified Outcome: Percentage of Patients With at Least 5% Weight Loss From Baseline at Week 24
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline body weight assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 220 | 217
percentage of participants | 3.2 | 5.1

9. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than 7% at Week 24
Description: The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 14 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 221 | 215
percentage of participants | 38.5 | 56.3

10. Secondary Outcome: Percentage of Patients With Glycosylated Hemoglobin (HbA1c) Level Less Than or Equal to 6.5% at Week 24
Description: as for outcome 9
Time Frame: Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 221 | 215
percentage of participants | 16.3 | 32.1

11. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy During the Double-blind Period
Description: Routine fasting SMPG, central laboratory FPG and HbA1c values were used to determine the requirement of rescue medication. If fasting SMPG value exceeded the specified limit for 3 consecutive days, the central laboratory FPG and HbA1c were performed. Threshold values - from baseline to Week 8: fasting SMPG/FPG >200 milligram/deciliter (mg/dL) (11.1 mmol/L) or HbA1c >9%, from Week 8 to Week 24: fasting SMPG/FPG >180 mg/dL (10.0 mmol/L) or HbA1c >8.5%. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 223 | 223
percentage of participants | 0.4 | 0.4

12. Secondary Outcome: Change From Baseline in Treatment Satisfaction Score (Sum of Items 1, 4, 5, 6, 7 and 8 of DTSQ) at Week 24
Description: Change was calculated by subtracting baseline value from Week 24 value. DTSQ: 8-item questionnaire to assess treatment satisfaction and patient perception of hyper and hypoglycemia. Each question (Q) scored on a Likert scale from 0 to 6. Six items (Q1 and 4-8; higher score = more satisfaction) measured treatment satisfaction and were summed to calculate treatment satisfaction score which ranged from 0 (very dissatisfied) to 36 (very satisfied). Two items (Q2 and 3), which were not included, measured perceived hyperglycemia and hypoglycemia, respectively and lower scores represented good perceived blood glucose control. The on-treatment period for this efficacy variable is the time from the first dose of study drug up to 3 days after the last dose of study drug or up to the introduction of rescue therapy, whichever is the earliest. For a patient to be included in mITT population, both baseline and at least 1 post baseline assessment for at least 1 efficacy variable, were required.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of patients analyzed = patients with baseline and at least 1 post-baseline DTSQ assessment during on-treatment period. Missing data was imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 209 | 201
units on a scale | 0.65 (0.545) | 0.88 (0.543)

13. Other Pre Specified Outcome: Number of Patients With Symptomatic Hypoglycemia and Severe Symptomatic Hypoglycemia
Description: Symptomatic hypoglycemia was an event with clinical symptoms that were considered to result from a hypoglycemic episode with an accompanying plasma glucose less than 60 mg/dL (3.3 mmol/L) or associated with prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration if no plasma glucose measurement was available. Severe symptomatic hypoglycemia was symptomatic hypoglycemia event in which the patient required the assistance of another person and was associated with either a plasma glucose level below 36 mg/dL (2.0 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, if no plasma glucose measurement was available.
Time Frame: First dose of study drug up to 3 days after the last dose administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Placebo | Lixisenatide
Number analyzed (Participants) | 223 | 223
participants
  Symptomatic hypoglycemia | 30 | 50
  Severe symptomatic hypoglycemia | 0 | 1

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 3 days after the last dose administration
Description: Median exposure to study treatment was 169 days in both treatment arms. The analysis was performed on safety population, defined as all randomized patients who were exposed to at least 1 dose of study drug, regardless of the amount of treatment administered.
Arm/Group | Placebo | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 10/223 | 17/223
Other Adverse Events (participants affected / at risk) | 81/223 | 127/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | Lixisenatide (N=223)
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=223) | Lixisenatide (N=223)
Influenza (Infections and infestations) | 14 | 11
Nasopharyngitis (Infections and infestations) | 12 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 43 | 61 — Hypoglycaemia adverse event is based on investigator reported hypoglycaemia.
Dizziness (Nervous system disorders) | 6 | 12
Headache (Nervous system disorders) | 8 | 22
Tremor (Nervous system disorders) | 4 | 13
Diarrhoea (Gastrointestinal disorders) | 7 | 15
Nausea (Gastrointestinal disorders) | 11 | 61
Vomiting (Gastrointestinal disorders) | 3 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.